CLINICAL TRIAL: NCT03746002
Title: Diuretic Effect of Metolazone Pre-dosing Versus Concurrent Dosing With Furosemide: a Pilot Study
Brief Title: Diuretic Effect of Metolazone Pre-dosing Versus Concurrent Dosing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient rate of patient enrollment/accrual.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Brent Reed, Associate Professor, Pharmacy Practice and Science, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00082982
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Fluid Overload; Heart Failure Acute
Keywords: diuretic; metolazone; furosemide
MeSH Terms: conditions — Edema | interventions — Metolazone; Furosemide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, active control pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metolazone Pre-dosing (Active Comparator): Metolazone 5 mg by mouth administered 60 minutes prior to furosemide background therapy (120 - 160 mg intravenous bolus, followed by furosemide 120 - 160 mg intravenous bolus 12 - 24 hours after)
  Interventions: Drug: Metolazone 60 minutes prior to furosemide
- Metolazone Concurrent Dosing (Active Comparator): Metolazone 5 mg by mouth administered at the same time as furosemide background therapy (120 - 160 mg intravenous bolus, followed by furosemide 120 - 160 mg intravenous bolus 12 - 24 hours after)
  Interventions: Drug: Metolazone concurrently with furosemide

INTERVENTIONS:
Drug: Metolazone 60 minutes prior to furosemide — All patients will receive furosemide background therapy (furosemide 120 - 160 mg IV bolus dosed twice within a twenty four hour period. Patients will be randomized 1:1 to either metolazone 5 mg tablet dosed 60 minutes prior to first dose of furosemide or metolazone dosed concurrently (within ten minute time frame) with the first dose of furosemide.
  Other Names: Zaroxolyn
  Arms: Metolazone Pre-dosing
Drug: Metolazone concurrently with furosemide — All patients will receive furosemide background therapy (furosemide 120 - 160 mg IV bolus dosed twice within a twenty four hour period. Patients will be randomized 1:1 to either metolazone 5 mg tablet dosed 60 minutes prior to first dose of furosemide or metolazone dosed concurrently (within ten minute time frame) with the first dose of furosemide.
  Other Names: Zaroxolyn
  Arms: Metolazone Concurrent Dosing

SUMMARY:
The purpose of this study is to examine whether administering metolazone 60 minutes prior to furosemide increases urine output compared with administering metolazone and furosemide concomitantly. Participants will have equal chance of being assigned to each group.

DETAILED DESCRIPTION:
Diuretic resistance is common among patients with acute decompensated heart failure, and one strategy for overcoming this phenomenon is sequential nephron blockade with loop plus thiazide-type diuretics. Metolazone is an oral thiazide-type diuretic commonly used for this purpose. Due to its delayed absorption, some clinicians suggest that metolazone be given 30-60 minutes prior to the loop diuretic. However, the efficacy and safety of such a strategy has not been investigated despite its added complexity. The purpose of this study is to investigate whether pre-dosing with metolazone confers a difference in efficacy and safety compared to administering it at the same time as furosemide.

ELIGIBILITY:
Inclusion Criteria:

* Admission within 48 hours for acute decompensated heart failure with at least one symptom and one sign of volume overload
* Receipt of loop diuretic prior to admission
* Plan to administer furosemide 120 - 160 mg IV bolus twice daily over the next 24 hours with additional diuresis deemed necessary
* If patient is concurrently administered intravenous vasodilator or inotrope, the dose of vasodilator or inotrope must be stable for 6 hours prior to enrollment with a plan to continue the same dose for the 24 hour duration of this study

Exclusion Criteria:

* Metolazone prescribed prior to admission
* Receipt of continuous intravenous infusion of furosemide
* Cirrhosis or end stage renal disease
* Non-English speaking patients

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Reed, PharmD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellison DH, Felker GM. Diuretic Treatment in Heart Failure. N Engl J Med. 2017 Nov 16;377(20):1964-1975. doi: 10.1056/NEJMra1703100. No abstract available. PMID 29141174
- [Background] Jentzer JC, DeWald TA, Hernandez AF. Combination of loop diuretics with thiazide-type diuretics in heart failure. J Am Coll Cardiol. 2010 Nov 2;56(19):1527-34. doi: 10.1016/j.jacc.2010.06.034. PMID 21029871
- [Background] Grosskopf I, Rabinovitz M, Rosenfeld JB. Combination of furosemide and metolazone in the treatment of severe congestive heart failure. Isr J Med Sci. 1986 Nov;22(11):787-90. PMID 3793436
- [Background] Ellison DH. The physiologic basis of diuretic synergism: its role in treating diuretic resistance. Ann Intern Med. 1991 May 15;114(10):886-94. doi: 10.7326/0003-4819-114-10-886. PMID 2014951

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metolazone Pre-dosing | Metolazone Concurrent Dosing
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metolazone Pre-dosing | Metolazone Concurrent Dosing | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (NA) — This group only had one participant so standard deviation does not apply. | 66 (7.1) | 57 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 50 (NA) — This group only had one participant so standard deviation does not apply. | 53 (10.6) | 51.7 (7.6)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1 (NA) — This group only had one participant so standard deviation does not apply. | 2.1 (0.6) | 1.8 (0.8)
Serum sodium [Mean (Standard Deviation); unit: mmol/L] | 138 (NA) — This group only had one participant so standard deviation does not apply. | 142 (6.4) | 140.3 (4.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 134 (NA) — This group only had one participant so standard deviation does not apply. | 132 (17) | 132.7 (12)
Total daily dose loop diuretic prior to admission (in oral furosemide equivalents) [Mean (Standard Deviation); unit: mg/day] | 100 (NA) — This group only had one participant so standard deviation does not apply. | 140 (28.3) | 126.7 (30.6)

OUTCOME MEASURES:

1. Primary Outcome: 24-Hour Urine Output
Description: Total measured urine output in milliliters produced after metolazone dose is given
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
mL | 2030 (1626.3) | 5650 (NA) — This group only had one participant so standard deviation does not apply.

2. Secondary Outcome: Change in Total Body Weight
Description: Change in total body weight from baseline value measured prior to metolazone dose to value collected after metolazone dose
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
kg | -.6 (1.1) | -8.5 (NA) — This group only had one participant so standard deviation does not apply.

3. Secondary Outcome: Change in Serum Creatinine
Description: Change in serum creatinine from baseline value collected prior to metolazone dose to value collected after metolazone dose
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
mg/dL | 0.45 (0.28) | 0.38 (NA) — This group only had one participant so standard deviation does not apply.

4. Secondary Outcome: Acute Kidney Injury
Description: Portion of patients with increase in serum creatinine by ≥ 0.3 mg/dL or ≥ 50% from baseline
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

5. Secondary Outcome: Hypokalemia
Description: Proportion of patients with potassium level less than 4.0 mEq/L measured after metolazone dose is given
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

6. Secondary Outcome: Hypomagnesemia
Description: Proportion of patients with magnesium level less than 2.0 mg/dL measured after metolazone dose is given
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

7. Secondary Outcome: Hyponatremia
Description: Proportion of patients with serum sodium level less than 135 mg/dL measured after metolazone dose is given
Time Frame: Baseline and at 12 to 23 hours after metolazone dose
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone Concurrent Dosing | Metolazone Pre-dosing
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours after metolazone dose (no greater than 48 hours after enrollment)
Arm/Group | Metolazone Pre-dosing | Metolazone Concurrent Dosing
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metolazone Pre-dosing (N=1) | Metolazone Concurrent Dosing (N=2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) — Defined as an increase in serum creatinine by 0.3 mg/dL or more, or 50% or more from baseline

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow enrollment, resulting in an inadequate sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03746002/Prot_SAP_001.pdf